CLINICAL TRIAL: NCT07201350
Title: The Impact on Fear and Anxiety Levels of Children of an Undersea-Themed Cover Designed for Electrocardiography Applications: A Randomized Controlled Trial
Brief Title: The Effect of an Undersea-Themed ECG Cover on Fear and Anxiety Levels in Children
Acronym: UTETC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, AYLİN ARIKAN, PhD, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UTETC
Record Dates: First submitted 2024-01-06; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Fear
Keywords: children; Pediatric ECG; Undersea-themed cover; Distraction technique; Pediatric emergency
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were stratified by age and gender, and then assigned to the intervention or control group using block randomization.
Who Masked: Outcomes Assessor
Masking Description: The outcomes were assessed by two independent nurses who were blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: distraciton technices
- Control (No Intervention)

INTERVENTIONS:
Other: distraciton technices — UTETC is a distraction method used during ECG procedures.
  Arms: Intervention

SUMMARY:
Aims: To evaluate the impact of an undersea-themed examination table cover (UTETC) designed for electrocardiography (ECG) procedures on fear and anxiety levels in children.

Background: Children may experience fear and anxiety not only during painful procedures but also during painless interventions such as ECG. The unfamiliar environment, equipment, and separation from caregivers can contribute to emotional distress.

Design: This is a single-blind, randomized controlled trial.

Methods: The study was conducted with 80 children aged 3-12 years who underwent ECG procedures in a pediatric emergency department. Participants were randomly assigned to either the control group (n = 40) or the intervention group (n = 40) using block randomization. Data were collected using the Child Fear Scale and the Children's Emotional Manifestation Scale.

Relevance to Clinical Practice: The UTETC represents a potential non-pharmacological intervention aimed at improving the emotional comfort of children during ECG procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 12 years
* Presented to the hospital with chest pain
* No previous history of heart disease
* Chest pain with a non-cardiac etiology (e.g., gastrointestinal disorders)
* Undergoing their first ECG

Exclusion Criteria:

-Reported fear of water, being underwater, or swimming

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
fear | 2 minutes before the ECG procedure, at the moment the ECG recording button is pressed, and 2 minutes after the ECG procedure
  Children's fear levels will be assessed using the Children's Fear Scale (CFS), which consists of five faces ranging from 0 (no fear) to 4 (extreme fear). Higher scores indicate higher levels of perceived fear.
anxiety | 2 minutes before the ECG procedure, at the moment the ECG recording button is pressed, and 2 minutes after the ECG procedure
  Anxiety will be assessed using the Children's Emotional Manifestation Scale (CEMS), which evaluates five categories of observable emotional behavior. Each item is scored from 1 to 5, with total scores ranging from 5 to 25. Higher scores indicate higher levels of observed anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- r Sami Ulus Maternity and Children's Health and Diseases Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No